CLINICAL TRIAL: NCT02892487
Title: Evaluation of an Active Swallowing Rehabilitation on Quality of Life of Patients Treated by Radiotherapy for Head and Neck Cancer
Acronym: RORC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For financial reasons and speed of recruitment was much slower than expected, inclusions weren't resumed after it was suspended during COVID-19 confinment.
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC14_9786_RORC
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cancer of Head and Neck
Keywords: Quality of life; Radiotherapy; Dysphagia; Oral cavity; Oropharynx; Hypopharynx; Larynx; Swallowing rehabilitation; Toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early active swallowing therapy (Experimental)
  Interventions: Other: Swallowing therapy
- Usual care (No Intervention)

INTERVENTIONS:
Other: Swallowing therapy — Patients will undergo active swallowing therapy with a speech and language therapist (twice a week) combined to a detailed program of swallowing auto-exercises (twice a day) from start of radiotherapy to one month after the end.
  Arms: Early active swallowing therapy

SUMMARY:
Toxicity and mainly dysphagia have increased in head and neck cancers as chemoradiation indications have risen over the last decade, leading to a significant loss of quality of life for patients. Recently, many retrospective studies and two evidence-based and systematic reviews on strategies to reduce radiation-induced dysphagia have suggested a trend toward benefit for a preventive swallowing exercise program.

The main hypothesis of this study is that an early active swallowing therapy can improve the Quality of Life (QoL) of patients treated by radiotherapy for head and neck cancer.

The study will be a randomized controlled, open-label, multicentric phase III clinical trial comparing early active swallowing therapy versus non specific swallowing management (usual care).

DETAILED DESCRIPTION:
Patients in both groups will receive dietary and postural advice from the treating physician. Patients in the experimental group will be treated with an early active swallowing therapy including a consultation with a speech and language therapist twice a week and a detailed program of swallowing auto-exercises twice a day, from the start to one month after the end of radiotherapy. All speech therapists will be given precise guidelines based on the current state of the art and knowledge. All patients will be analyzed in intent-to-treat.

Two ancillary studies will complete this global concept of the evaluation and prediction of severe alteration of Quality of Life (QoL) and Dysphagia.

1. A first study will evaluate videoradioscopy. Its objectives are to evaluate the ability of videoradioscopy at 3 months to predict poor QoL at 6 and 12 months, to identify videoradioscopic predictors of severe dysphagia, asymptomatic aspirations, cricopharyngeal stenoses and active swallowing rehabilitation efficiency. Each patient of both arms of the main study will undergo a videoradioscopy before the beginning of the radiation delivery (baseline evaluation), and at 3 and at 12 months. Data analysis will be centralized and will concern: APS (Aspiration and Penetration Scale) score, residue, Defective Laryngeal elevation, pharyngoesophageal sphincter dysfunction. Data will be correlated to the parameters of the main study in order to establish predictive models.
2. A second ancillary study will evaluate the dose-volume histograms of radiotherapy. The objectives are to identify predictors of dysphagia and of active swallowing rehabilitation efficiency, and to establish "2D" and "3D" predictive models of dysphagia. Imaging and dosimetric data (IMRT (Intensity Modified RadioTherapy) planning) and dose-volume histogram will be collected from the patients of the main clinical trial. Analysis will be centralized. Data will be correlated to the parameters of the main study in order to establish predictive models.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for histologically proven head and neck cancer (oral cavity, oropharynx, or hypopharynx cancer) of stages I-IV or larynx cancer of stages II-IV, all histologic type, without distant metastasis
* Indication of curative radiotherapy alone or associated to chemotherapy or targeted therapy, without planned surgery
* WHO (World Health Organization) Performance Status 0, 1 or 2
* Sufficient cognitive capacities to complete a QoL questionnaire (evaluation by the physician at inclusion)
* Written informed consent
* Patients with health insurance

Exclusion Criteria:

* Previous radiotherapy or surgery of the upper aerodigestive tract
* Cancer of paranasal sinuses or nasopharynx or skull base
* Medical history of nervous system disease associated to significant sequelae in terms of dysphagia
* Pregnant or breast-feeding woman
* Patient under guardianship, trusteeship or judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing a clinically relevant improvement defined as a decrease of at least 10 points of the score HNSW ( 6 months after radiotherapy compared with the score before radiotherapy | 6 months after radiotherapy
  HNSW = Head and Neck Swallowing Questionnaire

SECONDARY OUTCOMES:
EORTC QLQ-C30 score | Baseline, 3, 6 and 12 months after radiotherapy
  EORTC QLQ = European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire
EORTC H&N35 score | Baseline, 3, 6 and 12 months after radiotherapy
  EORTC H&N = European Organisation for Research and Treatment of Cancer Head and Neck questionnaire
MFI-20 score | Baseline, 3, 6 and 12 months after radiotherapy
  MFI = Multidimensional Fatigue Inventory
Body Mass index (BMI) | Baseline, 3, 6 and 12 months after radiotherapy
  in kg/m^2
Functional Oral Intake Scale (FOIS) | Baseline, 3, 6 and 12 months after radiotherapy
Overall duration of enteral nutrition | 12 months after radiotherapy
Total treatment duration | 12 months after radiotherapy
Number of treatment interruptions | 12 months after radiotherapy
Number of patients with adverse events | End of radiotherapy (an average of 2 months after baseline), 1, 3, 6 and 12 months after radiotherapy
Swallowing specific Quality of Life (SWAL-QOL) score | Baseline, 3, 6 and 12 months after radiotherapy
Number of patients with aspiration and penetration determined by APS (Aspiration and Penetration Scale) scoring | Baseline, 3, 6 and 12 months after radiotherapy
Rate of global survival | 12 months after radiotherapy
Rate of survival without recurrence | 12 months after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Franck JEGOUX, Principal Investigator — Rennes University Hospital
Locations (21):
- France (21):
  - Brest University Hospital, Brest
  - Caen University Hospital, Caen
  - Centre François Baclesse, Caen
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Le Mans Hospital, Le Mans
  - Lille University Hospital, Lille
  - Bretagne Sud Hospital, Lorient
  - Lyon University Hospital, Lyon
  - Marseille University Hospital, Marseille
  - Centre Alexis Vautrin, Nancy
  - Nantes University Hospital, Nantes
  - Centre Antoine Lacassagne, Nice
  - Tenon Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Clinique La Sagesse, Rennes
  - Rennes University Hospital, Rennes
  - Strasbourg University Hospital, Strasbourg
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours
  - Bretagne Atlantique Hospital, Vannes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No